CLINICAL TRIAL: NCT06921200
Title: Effect of Perineal Cryotherapy on Episiotomy- Associated Pain Among Postpartum Women
Brief Title: Effect of Perineal Cryotherapy on Episiotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Ahmed Fadel, Assistant professor of Woman's Health and Midwifery Nursing, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB. 0562
Record Dates: First submitted 2025-03-03; First posted 2025-04-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-02

CONDITIONS: Normal Vaginal Delivery; Perineal Episiotomy
Keywords: Episiotomy; Pain; Perineal cryotherapy
MeSH Terms: conditions — Pain | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-partum women who apply perineal cryotherapy after normal vaginal delivery with episiotomy (Experimental): Apply perineal cryotherapy after normal vaginal delivery with episiotomy (interventional group)
  Interventions: Procedure: Cryotherapy
- control group (No Intervention): Postpartum women who receive routine episiotomy care after normal delivery

INTERVENTIONS:
Procedure: Cryotherapy — Cryotherapy is one of the non-pharmacological pain-relieving techniques, which involves chilling specific body areas with ice packs, ice cubes, ice water, or ethyl chloride sprays. The present study intervention will be conducted on 50 post-partum women to assist in relieve episiotomy pain. The researchers will assess the baseline level of episiotomy pain for each woman then the researchers will instruct women to perform perineal care. After cleaning the perineum, the researchers will ask the women to maintain her knee more flexed and apply ice gel pad against the episiotomy line for about 20 minutes then remove it and keep it in the freezer for reusing and assess the level of episiotomy pain using the Numeric Rating Scale for Pain after two hours from delivery. Ice gel pad will be applied for the second time after the episiotomy.
  Arms: Post-partum women who apply perineal cryotherapy after normal vaginal delivery with episiotomy

SUMMARY:
The present study aims to evaluate the effect of perineal cryotherapy on episiotomy- associated pain among postpartum women.

The study hypothesis: Post-partum women who apply perineal cryotherapy have lower level of episiotomy- associated pain than those who don't apply.

DETAILED DESCRIPTION:
The present study included postpartum mothers who are in a good health immediately after giving delivery, having an episiotomy and a normal vaginal birth of a single, full term, healthy baby with normal weight and vertex presentation.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum mothers who are in a good health immediately after giving delivery.
* Having an episiotomy and a normal vaginal birth.
* Having a vaginal birth at full term.
* The delivery of a healthy single fetus having normal weight and vertex presentation.

Exclusion Criteria:

* Women who are experiencing labor or complications after giving birth, such as hemorrhage, a tear, or a cut in the perineum.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Level of episiotomy-associated pain | from enrollmet until four hours after delivery